CLINICAL TRIAL: NCT07357285
Title: Prospective, Single-arm, Multi-centre Study to Evaluate the Efficacy and Safety of the iNstroke 4F Thromboaspiration Catheter in Patients With Acute Ischaemic Stroke Due to Primary Distal Medium Vessel Occlusions (DMVO).
Brief Title: Safety and Efficacy Evaluation of the iNstroke 4F Thromboaspiration Catheter in Patients With Acute Ischaemic Stroke Due to Primary Distal Medium Vessel Occlusions (DMVO)
Acronym: 4-NiVO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: iVascular S.L.U. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-NiVO-01
Record Dates: First submitted 2025-12-09; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Ischemia; Thromboaspiration
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thromboaspiration using iNstroke 4F aspiration catheter (Other): No comparator will be used in this clinical investigation as it is an exploratory study of a CE-marked medical device to be used within the scope of its intended purpose.
  Interventions: Device: Thromboaspiration catheter

INTERVENTIONS:
Device: Thromboaspiration catheter — Patients to undergo thromboaspiration with iNstroke 4F

SUMMARY:
Prospective, Single-arm, Multi-centre Study to Evaluate the Efficacy and Safety of the iNstroke 4F Thromboaspiration Catheter in Patients with Acute Ischaemic Stroke due to Primary Distal Medium Vessel Occlusions.

DETAILED DESCRIPTION:
This study is an exploratory, interventional, open label, single-arm, multi-centre prospective clinical investigation.

In this post-market clinical investigation, the aim is to further evaluate the efficacy and safety of the iNstroke 4F aspiration catheter, with a view to, in future clinical investigations, comparing the product with the standard therapy or with other similar products. In addition, this clinical investigation will generate results that could be used to further assess the safety and effectiveness of mechanical thrombectomy for the treatment of DMVO.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 years.
* Subjects with symptom onset up to 24 hours.
* Isolated primary demonstrated occlusion in a distal medium vessel (Non-dominant or distal M2-MCA segment, M3 or M4 segments of MCA, A2-A3 segments of ACA, P1, P2 and P3 segments of PCA) identified by magnetic resonance angiography (MRA) or computed tomography angiography (CTA).
* Baseline NIHSS score ≥5 assessed before the procedure.
* Pre-stroke mRS score ≤ 2.
* Subjects with an ASPECTS score ≥ 6.
* Informed consent obtained in accordance with the applicable country-specific regulations and as approved by the Ethics Committee (EC).

Exclusion Criteria:

* Subjects aged < 18.
* Suspected secondary DMVO. Suspicion or evidence of primary LVO whether it has been treated or not with fibrinolytic therapy or mechanical thrombectomy that subsequently develops a DMVO.
* Baseline NIHSS score <5 assessed before the procedure.
* Pre-stroke mRS score >2.
* Subjects with an ASPECTS score <6.
* Severe comorbidity and/or shortened life expectancy that will likely prevent improvement or follow up or that will render the procedure unlikely to benefit the patient.
* Severe allergy to contrast media.
* Subjects with intracranial atherosclerotic occlusive disease or extra- or intracranial dissection.
* Medical history of thrombocytopenia (Platelets <100,000).
* Subjects with tandem occlusions (evidence of complete occlusion, high-grade stenosis or arterial dissection in the extracranial or petrous segment of the internal carotid artery).
* Subjects with occlusions in multiple vessels (e.g., MCA-M3 and ACA-A2), whether or not they undergo mechanical thrombectomy.
* Subjects with cancer (with or without metastases) who have a life expectancy of less than 6 months.
* Subjects participating in a clinical trial at the moment of the inclusion.
* Subjects with pre-existing neurological or psychiatric illness that could confound the neurological or functional assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Recanalization Endpoint | Intra-procedure
  Recanalization rate with a modified thrombolysis in cerebral infarction scale (mTICI) score ≥2b in ≤3 revascularization passes using iNstroke 4F aspiration catheter, alone or in conjunction with a SR.

SECONDARY OUTCOMES:
Recanalization Endpoint | Intra-procedure
  Proportion of subjects treated with iNstroke 4F alone with complete recanalization in primary DMVO defined as an mTICI ≥2b, after iNstroke 4F aspiration catheter alone (ADAPT) was used as a first-line therapy
Recanalization Endpoint | Intra-procedure
  Proportion of subjects treated with iNstroke 4F in conjunction with a stent retriever having complete recanalization in primary DMVO defined as achieving an mTICI ≥2b, after iNstroke 4F aspiration catheter, in conjunction with a stent retriever (SR), was used as a first-line therapy.
Recanalization Endpoint | Intra-procedure
  Proportion of subjects with mTICI≥2b, mTICI≥2c and mTICI 3 after first pass with iNstroke 4F aspiration catheter used both alone and in conjunction with a SR.
Recanalization Endpoint | Intra-procedure
  Time from groin puncture to achievement of complete recanalization (mTICI ≥2b), or if not achieved, until the final angiogram time, in patients treated with iNstroke 4F aspiration catheter, alone or in conjunction with a SR, as a first-line therapy.
Recanalization Endpoint | Intra-procedure
  Proportion of subjects in which direct contact with thrombus is achieved with iNstroke 4F aspiration catheter.
Clinical Endpoint | 90 day
  Proportion of subjects achieving a modified Rankin scale (mRS) score of 0-2 at the 90-day (±14 days) post-procedure follow-up visit.
Safety Endpoint | 24 (-8/+12) hours
  Occurrence of SICH (according to SITS-MOST (13) and ECASS criteria (14)) within 24 (-8/+12) hours post-procedure, assessed by magnetic resonance imaging (MRI)/computed tomography (CT).
  Intracerebral Haemorrhage (ICH) is defined as the presence of extravascular blood in the brain or within the skull (local or remote parenchymal hematoma type 2, subarachnoid haemorrhage, and/or intraventricular haemorrhage) detected on the post-procedure imaging scan. ICH is considered symptomatic (SICH) if it is associated with a clinical deterioration, determined by a worsening/increase on the National Institutes of Health Stroke Scale (NIHSS) score of ≥4 points, or if it causes death and is identified as the predominant cause of neurological deterioration.
Safety Endpoint | Intra-procedure
  Occurrence of embolization in a previously non-involved (or new) territory as seen on the final control angiogram at the end of the procedure.
Safety Endpoint | Intra-procedure
  Occurrence of embolization in distal medium territory to the proximal occlusion as seen on the final control angiogram at the end of the procedure.
Safety Endpoint | During hospital admission
  Inhospital mortality rate related to the procedure during hospital admission.
Safety Endpoint | 90 days (±14 days) after the procedure.
  Occurrence of devices and procedure related adverse events within 90 days (±14 days) after the procedure.
Safety Endpoint | Intra-procedure
  Occurrence of procedure-related complications: arterial perforation, arterial dissection and severe vasospasm in the target vessel.

OTHER OUTCOMES:
Exploratory Recanalization Endpoint | Intra-procedure
  Proportion of subjects in which a switch of technique (from ADAPT to combined or from combined to ADAPT) with iNstroke 4F aspiration catheter was used to successfully perform the thrombectomy.
Exploratory Recanalization Endpoint | Intra-procedure
  Proportion of subjects in which an aspiration catheter device with a 4F caliber different from iNstroke 4F aspiration catheter was used as a rescue therapy.
Exploratory Recanalization Endpoint | Intra-procedure
  Proportion of cases in which iNstroke 4F aspiration catheter (alone or in conjunction with a SR) successfully reached the site of occlusion.
Exploratory Recanalization Endpoint | Intra-procedure
  Number of passes with iNstroke 4F aspiration catheter until recanalization.
Exploratory Recanalization Endpoint | Intra-procedure
  Visibility of the catheter during the thrombectomy rated from 0 to 5 (being 0 the worst and 5 the best score).
Exploratory Clinical Endpoint | 24 (-8/+12) hours post-procedure.
  Proportion of subjects with rapid neurological improvement, defined as a decrease of more than 4 points on the NIHSS scale, during the first 24 (-8/+12) hours post-procedure.
Exploratory Clinical Endpoint | First 24 (-8/+12) hours post-procedure or 3 days (±24 hours) or at the time of discharge, whichever occurs first.
  Proportion of subjects with a reduction of ≥8 points on the NIHSS scale during the first 24 (-8/+12) hours post-procedure, or with a NIHSS score of 0-1 at 3 days (±24 hours) or at the time of discharge, whichever occurs first.
Exploratory Clinical Endpoint | 24 (-8/+12) hours.
  Median of NIHSS score at 24 (-8/+12) hours.
Exploratory Clinical Endpoint | 3 days (±24 hours) post procedure
  Median of NIHSS score at 3 days (±24 hours) or at the time of patient discharge, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (11):
- Germany (5):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Klinikum Marburg, Marburg
  - Klinikum Nürnberg, Nuremberg
  - Knappschaftskrankenhaus Recklinghausen, Recklinghausen
- Semmelweis University Center, Budapest, Hungary
- Spain (5):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Getafe, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario Virgen de Arrixaca, Murcia

IPD SHARING:
Plan to Share IPD: No